CLINICAL TRIAL: NCT03719911
Title: Evaluation of the Effects of a Technologically-Enhanced Personal Coaching Program on Hemoglobin A1c in Type 2 Diabetics
Brief Title: Evaluating the Impact of a Technologically-Enhanced Personal Coaching Program on Hemoglobin A1c in Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Welkin Health (Other)
Collaborators: LifeScan (Industry)
Responsible Party: Principal Investigator, Kristin Neland, Clinical Program Designer, Welkin Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTR_COACHING1
Record Dates: First submitted 2018-09-25; First posted 2018-10-25 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: single-arm 24-week pre-post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Live diabetes coaching program (Experimental): Live diabetes coaching program
  Interventions: Behavioral: Live diabetes coaching program

INTERVENTIONS:
Behavioral: Live diabetes coaching program — Live diabetes coaching program

SUMMARY:
Participants diagnosed with Type 2 diabetes receive personal coaching from a Certified Diabetic Educator (CDE) over a six-month period. The coaching program is enhanced using an mobile application and care management platform.

DETAILED DESCRIPTION:
Participants diagnosed with Type 2 diabetes receive personal coaching from a Certified Diabetic Educator (CDE) over a six-month period. The coaching program is enhanced by integrating a participant-facing mobile application with the coaching platform. Blood glucose test results automatically populate the coaching platform, providing the CDE with information that may better support their coaching efforts.

The participants complete Diabetes Self Management Education (DSME) learning modules for the first 7-12 weeks. Following completion of the modules, the coach continues to provide support to the participant until 24 weeks after the participant's enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Lives in the United States
* Speaks and understands English
* Has a Type 2 diabetes mellitus diagnosis
* Has a LifeScan Verio Flex blood glucose meter, which is connected to OneTouch Reveal ® app
* Has a verified A1c ≥ 8%
* Willing to participate in coaching program

Exclusion Criteria:

* Uses a continuous glucose monitoring device
* Currently pregnant
* Unable to make lifestyle behavioral changes due to a cognitive or physical disability
* Has end stage renal disease (ESRD) diagnosis
* Is not able to read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | A1c measured at baseline, at 12 weeks since study enrollment, and at 24 weeks since enrollment, which marks the participant's completion of the study
  Blood serum test to measure glucose control

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Neland, BSN, MPH, Principal Investigator — Welkin Health
Locations (1):
- Welkin Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Investigators will not share IPD with other researchers